CLINICAL TRIAL: NCT03284502
Title: A Phase Ib, Open-label, Multicenter, Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of HM95573 in Combination With Either Cobimetinib or Cetuximab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: HM95573 in Combination With Either Cobimetinib or Cetuximab in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-RAFI-103
Record Dates: First submitted 2017-08-07; First posted 2017-09-15 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Belvarafenib; HM95573; GDC-5573; RG6185; Cobimetinib; Cetuximab
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cobimetinib; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1 (Experimental): Dose-escalation
  Interventions: Drug: HM95573, cobimetinib
- Stage 1b (Experimental): Dose-escalation
  Interventions: Drug: HM95573, cetuximab
- Stage 2 (Cohort I and II) (Experimental): Dose-expansion
  Interventions: Drug: HM95573, cobimetinib
- Stage 2 (Cohort III) (Experimental): Dose-expansion
  Interventions: Drug: HM95573, cetuximab

INTERVENTIONS:
Drug: HM95573, cobimetinib — Regimen: twice daily (BID), continuous dosing for HM95573, once daily (QD) 21 days, 7 days off for cobimetinib
  Arms: Stage 1
Drug: HM95573, cetuximab — Regimen: twice daily (BID), continuous dosing for HM95573
  Arms: Stage 1b
Drug: HM95573, cobimetinib — Regimen: Recommended dose (RD) and schedule selected based on the data of safety, tolerability, pharmacokinetics, and anti-tumor activity tested in Stage 1
  Arms: Stage 2 (Cohort I and II)
Drug: HM95573, cetuximab — Regimen: Expansion dose of HM95573 selected based on the data of safety and tolerability tested in Stage 1b
  Arms: Stage 2 (Cohort III)

SUMMARY:
This study evaluates the safety, tolerability and pharmacokinetics of HM95573 In combination with either cobimetinib or cetuximab in patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a Phase Ib, open-label, multicenter dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of oral dosing of HM95573 in combination with either cobimetinib or cetuximab in patients with histologically/cytologically confirmed, locally advanced, or metastatic solid tumors with RAS- or RAF-mutation for which standard therapies either do not exist or have proven ineffective or intolerable. Treatment will continue until disease progression, unacceptable toxicity, any other discontinuation criterion is met.

There are two stages of this study: Stage 1 and 1b, standard 3+3 dose escalation, and Stage 2, an indication-specific dose expansion. Stage 1 is designed to establish the combination MTD for cobimetinib and HM95573. Stage 1 consists of concurrent administration of cobimetinib and HM95573. Stage 1b, is designed to select the combination dose of cetuximab and HM95573 for expansion stage.

In Stage 2 expansion cohort I and II, the RD of cobimetinib and HM95573 with different dosing schedules or regimens might be investigated (which may be≤ MTDs established during dose escalation) in indication-specific expansion cohorts. Stage 2 expansion cohort III will further characterize the safety and tolerability of cetuximab in combination with HM95573.

ELIGIBILITY:
[Inclusion criteria]

1. Signed Informed Consent Form
2. Age ≥ 19 years at time of signing Informed Consent Form
3. ECOG performance status of 0 or 1
4. Histologically or cytologically documented, locally advanced or metastatic solid tumors with RAS- or RAF-mutation for which standard therapy either does not exist or has proven ineffective or intolerable
5. Measurable disease per RECIST v1.1
6. Life expectancy ≥ 12 weeks
7. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 2 weeks prior to the first dose of study-drug treatment: Absolute neutrophil count ≥ 1,500/μL Platelet count ≥ 100,000/μL Hemoglobin ≥ 9.0 g/dL (this criterion has to be met without transfusion within 2 weeks prior to laboratory test) Albumin ≥ 2.5 g/dL Total bilirubin ≤ 1.5 × ULN AST or ALT ≤ 3 × ULN, ALP ≤ 2.5 × ULN, with the following exceptions:

   * Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN
   * Patients with documented liver or bone metastases:

   ALP ≤ 5 × ULN Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min on the basis of the Cockroft-Gault glomerular filtration rate estimation PT/INR and PTT ≤ 1.5 × ULN
8. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use one highly effective form (defined as a failure rate of less than 1% per year) of contraception (e.g., surgical sterilization, birth control pills, or contraceptive hormone implants) and to continue use for the duration of the study. Additionally, female patients of childbearing potential should use pregnancy prevention measures for a minimum of 3 months following discontinuation of HM95573 in combination with either cobimetinib or cetuximab.
9. For male patients: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: For men with female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 3 months after the last dose of HM95573 in combination with either cobimetinib or cetuximab to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The length of time that pregnancy preventative measures are used following discontinuation of drug may be adjusted based on the human pharmacokinetics.
10. Consent to provide archival tissue (either a paraffin-embedded tissue block or unstained slides) for testing with the FoundationOne panel to assess and confirm genetic alterations including, but not limited to, KRAS, NRAS, BRAF, EGFR and PI3K mutational status.
11. FDG-PET avid disease on baseline scan. Patients who are considered for enrollment into the cohort expansion (Stage 2) must meet all of the following additional eligibility criteria:
12. No more than five prior systemic therapies for locally advanced or metastatic cancer
13. For the expansion cohorts (except basket cohort in expansion cohort I, II): No prior therapy with a RAF, MEK or ERK inhibitor. No prior treatment with regorafenib in the CRC (KRAS G13D- and BRAF V600-mutant) expansion cohort II. No prior therapy with HM95573 or cobimetinib in the expansion cohort II. For Stage 1b and the expansion cohort III prior EGFR, RAF, MEK, ERK inhibitor is allowed.
14. Current cancer must be one of the following:

    * Expansion cohort I (HM95573 200 mg BID + cobimetinib 20 mg QD):

      * KRAS-mutant NSCLC
      * KRAS-mutant Pancreatic adenocarcinoma
      * RAS-mutant CRC
      * RAS- or RAF-mutant solid tumors (basket cohort; excludes KRAS-mutant NSCLC, KRAS-mutant pancreatic adenocarcinoma, and RAS-mutant CRC). A minimum of 10 melanoma patients will be enrolled.
    * Expansion cohort II (HM95573 300 mg BID + cobimetinib 20mg QOD (3 times a week: day 1, 3, 5, 8, 10, 12, 15, 17, 19 of 28 day cycle)):

      * KRAS G13D-mutant CRC
      * BRAF V600-mutant CRC
      * NRAS-mutant Melanoma
      * RAS- or RAF-mutant solid tumors (basket cohort: A minimum of 10 BRAF V600 melanoma will be enrolled)
      * BRAF Class II-mutant (including BRAF fusions) or Class IIImutant solid tumors
    * Stage 1b and Expansion cohort III (HM95573 selected dose from stage 1b + cetuximab): - BRAF V600-mutant CRC
15. At least one target lesion on CT must also be an FDG-PET avid region of interest which has a target-to-organ-background SUVmax (or similar radioactivity concentration measure) ratio of ≥ 2.0 and at least 15mm in longest diameter.
16. Consent to undergo pre- and post-treatment tumor biopsies for PD biomarker analysis is optional, provided sites of disease are easily and safely accessible. In the absence of easily and safely accessible sites of disease, patients may enroll without consenting to tumor biopsies (Stage 2).
17. Willingness to take prophylactic antibiotics and topical steroids for the management of skin toxicity unless otherwise contraindicated for patient in Stage 1b and Expansion cohort III.

[Exclusion criteria]

Patients who meet any of the following criteria will be excluded from study entry:

1. History of prior significant toxicity from another RAF, MEK, ERK, or EGFR inhibitor requiring discontinuation of treatment
2. History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for central serous retinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration. Patients will be excluded from study participation if they currently are known to have any of the following risk factors for RVO:

   * Grade ≥ 2 or symptomatic hyperglycemia (fasting)
   * Grade ≥ 2 uncontrolled hypertension (patients with a history of hypertension controlled with anti-hypertensive medication to Grade ≤ 1 are eligible)
3. History of glaucoma
4. Allergy or hypersensitivity to components of the cobimetinib, cetuximab or HM95573 formulation
5. Palliative radiotherapy within 2 weeks prior to first dose of study-drug treatment in Cycle 1
6. Experimental therapy within 4 weeks prior to first dose of study-drug treatment in Cycle 1
7. Major surgical procedure or significant traumatic injury within 4 weeks prior to the first dose of study-drug treatment in Cycle 1, or anticipation of the need for major surgery during the course of study treatment
8. Anti-cancer therapy within 28 days prior to the first dose of study-drug treatment in Cycle 1. Exceptions include a washout period of at least five half-lives for anti-PD1 or anti-PDL1 antibodies and ipilimumab during Stage I dose escalation and at least three halflives for anti-PD1 or anti-PDL1 antibodies and ipilimumab during Stage II expansion phase, a washout of 6 weeks for nitrosoureas or mitomycin C, or 14 days for hormonal therapy or kinase inhibitors. (upon discussion with the Medical Monitor, fewer than stated wash-out period may be allowed provided that the patient has adequately recovered from any clinically relevant toxicity).
9. Current Grade > 1 toxicity (except alopecia and anorexia) from prior therapy or Grade > 1 neuropathy from any cause
10. Current severe, uncontrolled systemic disease (including, but not limited to, clinically significant cardiovascular, pulmonary, or renal disease, ongoing or active infection)
11. History of clinically significant cardiac dysfunction, including the following: Current uncontrolled Grade ≥ 2 hypertension or unstable angina
12. History of symptomatic congestive heart failure of New York Heart Association class III or IV or serious cardiac arrhythmia requiring treatment, with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia
13. History of myocardial infarction within 6 months prior to the first dose of study-drug treatment in Cycle 1
14. History of bradyarrhythmias, bradycardia or heart block or baseline HR < 55bpm
15. History of congenital long QT syndrome or QTcF > 440 msec
16. LVEF (as measured by echocardiography [ECHO] or multi-plegated acquisition scan [MUGA]) < 50% or below the lower limit of normal (LLN; whichever is lower)
17. Inability or unwillingness to swallow pills
18. History of malabsorption or other condition that would interfere with enteral absorption
19. Clinically significant history of liver disease (including cirrhosis), current alcohol abuse, or current known active infection with HIV, hepatitis B virus, or hepatitis C virus
20. Any hemorrhage or bleeding event CTCAE Grade 3 or higher within 28 days of Cycle 1, Day 1
21. Patients receiving therapeutic anticoagulation or thrombolytic anticoagulants. Use of low molecular weight heparin and low dose aspirin are allowed.
22. Active autoimmune disease
23. Uncontrolled ascites requiring weekly large volume paracentesis for 3 consecutive weeks prior to enrollment
24. Pregnancy, lactation, or breastfeeding
25. Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms

    - Patients with a history of adequately treated brain metastases are eligible. Adequately treated brain metastases are defined as those having no ongoing requirement for medical therapy to control symptoms, and no evidence of progression or hemorrhage for ≥ 2 months after radiation treatment (such as whole brain radiotherapy or radiosurgery [Gamma Knife, linear accelerator, or equivalent]) and/or ≥ 3 months after surgical treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or CT scan) during the screening period. Any medical therapy for brain metastases (e.g., steroids or seizure medications) must have been discontinued without the subsequent appearance of symptoms for ≥ 4 weeks before the first dose of study-drug treatment in Cycle 1.
26. Inability to comply with study and follow-up procedures
27. No other history of or ongoing malignancy that would potentially interfere with the interpretation of the pharmacodynamics (PD) or efficacy assays
28. Need to take a concomitant medication, dietary supplement, or food that is prohibited during the study
29. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest as assessed by CTCAE v4.03 | up to approximately 3 years
Number of patients with DLTs | 28 days
MTDs of HM95573 and cobimetinib, or HM95573 and cetuximab | End of Stage 1, an approximately 2 years
Recommended Phase II dose (RPIID) of HM95573 and cobimetinib, or HM95573 and cetuximab | End of Stage 1, an approximately 2 years

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of HM95573 and cobimetinib, or HM95573 and cetuximab | Cycle1 Day1, Cycle1 Day15, Cycle1 Day21, Cycle2 Day1, Cycle3 Day1, Study completion, an approximately 2 years
Maximum Serum Concentration (Cmax) of HM95573 and cobimetinib, or HM95573 and cetuximab | Cycle1 Day1, Cycle1 Day15, Cycle1 Day21, Cycle2 Day1, Cycle3 Day1, Study completion, an approximately 2 years
Time to maximum concentration (Tmax) of HM95573 and cobimetinib, or HM95573 and cetuximab | Cycle1 Day1, Cycle1 Day15, Cycle1 Day21, Cycle2 Day1, Cycle3 Day1, Study completion, an approximately 2 years
FDG-PET and molecular biomarkers assessed in pre- and post-treatment tumor tissues | Screening, Cycle1 Day15
Preliminary assessment of the antitumor activity of HM95573 and cobimetinib, or HM95573 and cetuximab measured by RECIST v1.1. | Screening, During Days 22-28 (Day 25 ± 3 days) in Cycle 2 and 4, and then every 8 weeks (±7 days), until disease progression, assessed approximately 3 years

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Dong-A University Hospital, Pusan
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Borame Hospital, Seoul